CLINICAL TRIAL: NCT03308292
Title: Effects of Exercise in Different Sport Surfaces, Diet and Lifestyle in the Bone Density of Pre and Post Menopausal Women
Brief Title: Effects of an Exercise Program on Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, ÁLVARO FERNÁNDEZ LUNA, Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2016/UEM33
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Bone Density; Body Composition
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental): A moderate-intensity aerobic physical exercise programme was carried out during the months of March to May 2017 (12 weeks), with a frequency of three sessions per week (36 sessions in total) with a duration of 45 minutes per session. The intensity was controlled through the Borg 1982 modified scale of perceived exertion (RPE). It is a scale from 0 to 10, considering 0 as "nothing at all" and 10 as "very very strong", setting the moderate intensity as value
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Aerobic exercise program
  Arms: Intervention Group

SUMMARY:
Physical inactivity and low adherence to the Mediterranean diet cause alterations in body composition, which increases the risk factors for cardiovascular and metabolic diseases. In addition, exercise in different surfaces or water could affect the bone density specially in women. Objective: The purpose of the study was to analyze the effect of a short-term aerobic exercise program in different surfaces on the body composition and bone density of women within at work, and to evaluate the quality of the Mediterranean diet and distribution of macronutrients in the studied population. Material & Methods: Randomized controlled trial. 63 women from a randomized work environment (IG, n=34) and a control group (CG, n=29) participated in a short-term aerobic exercise programmed (12 weeks), for body composition and bone density Dual-energy X-ray absorptiometry (DXA) was used and to evaluate diet, the Mediterranean Diet Quality Questionnaire (KIDMED) and the Food Frequency Questionnaire for macronutrient distribution were used.

ELIGIBILITY:
Inclusion Criteria:

* Not diagnosed with any disease that contraindicates the practice of physical exercise
* Do not perform physical activity with continuity

Exclusion Criteria:

* Diagnosed with chronic disease including cardiovascular and respiratory diseases that contraindicate the practice of physical exercise
* Being pregnant before or during the intervention (for intervention and control group)

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Changes in bone density | 3 months
  Change from baseline to 3 months using Dual-energy X-ray Absorptiometry
Changes in body composition | 3 months
  Change from baseline to 3 months using Dual-energy X-ray Absorptiometry

SECONDARY OUTCOMES:
Level of compliance with the exercise program | 3 months
  Level of compliance with the program using the percentage of compliance to the exercise programme (36 sessions)
Changes in Dietary pattern variables: macronutrients | 3 months
  Evaluation of Changes in Dietary pattern variables from baseline to 3 months using questionaries
Changes in Dietary pattern variables: quality of diet | 3 months
  Evaluation of Changes in Dietary pattern variables from baseline to 3 months using questionaries

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iturriaga T, Barcelo O, Diez-Vega I, Cordero J, Pulgar S, Fernandez-Luna A, Perez-Ruiz M. Effects of a short workplace exercise program on body composition in women: A randomized controlled trial. Health Care Women Int. 2020 Feb;41(2):133-146. doi: 10.1080/07399332.2019.1679813. Epub 2019 Oct 22. PMID 31638477